CLINICAL TRIAL: NCT04072250
Title: Surgery for Recurrent Intrahepatic Cholangiocarcinoma: a Promise or an Excess?
Brief Title: Surgery for Recurrent Intrahepatic Cholangiocarcinoma
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201701127B0
Record Dates: First submitted 2019-08-26; First posted 2019-08-28 (Actual); Last update posted 2019-09-13 (Actual); Status verified 2018-01

CONDITIONS: Cholangiocarcinoma, Intrahepatic; Recurrence Cholangiocarcinoma; Re-hepatectomy
Keywords: Recurrent intrahepatic cholangiocarcinoma; Intrahepatic cholangiocarcinoma; Repeat hepatectomy; Metastasectomy
MeSH Terms: conditions — Cholangiocarcinoma | interventions — Hepatectomy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: hepatectomy — Hepatectomy for patients with recurrent intrahepatic cholanigocarcinoma

SUMMARY:
The investigators retrospectively reviewed the participants suffering from recurrent intrahepatic cholangiocarcinoma after curative resection and aimed to explore the predictive factors for recurrence and clarify the potential benefit of repeat hepatectomy or/with metastasectomy.

ELIGIBILITY:
Inclusion Criteria:

* R0 resection for intrahepatic cholangiocarcinoma at initial diagnosis.

Exclusion Criteria:

* (1)Patient with R1 or R2 resection
* (2)Distant metastasis noted when laparotomy
* (3)Surgical mortality

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Between January 1977 and December 2014, 452 patients underwent curative-intent, different extent of hepatectomy for ICC in the Department of General Surgery, Chang Gung Memorial Hospital, Linkou branch, Taiwan. Only 216 patients fulfilled selection criteria aforementioned.
Sampling Method: Non-Probability Sample
Enrollment: 216 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2018-10-30 (Actual)

PRIMARY OUTCOMES:
Survival | 1977~2014
  Including overall survival and disease free survival

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memorial Hospital Linkou Branch, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No